CLINICAL TRIAL: NCT06965231
Title: Efficacy and Safety of Perioperative Toripalimab Combined With Recombinant Human Endostatin as Postoperative Adjuvant Therapy for Clinical Stage II Malignant Melanoma: A Multicenter, Single-Arm, Phase II Clinical Study
Brief Title: Perioperative Toripalimab and Endostatin for Stage II Melanoma: A Phase II Trial
Acronym: FUMS-EDJS2024
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: Shanghai Tongren Hospital, Shanghai Jiao Tong University School of Medicine (Unknown); Shanghai 411 hospital (Unknown)
Responsible Party: Principal Investigator, Chunmeng Wang, Director, Head of Musculoskeletal Oncology, Principal Investigator, Clinical Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB2501312-12
Record Dates: First submitted 2025-04-18; First posted 2025-05-11 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Melanoma of Skin; Acral Melanoma; Stage II Melanoma
Keywords: Melanoma of skin; Acral melanoma; Stage II melanoma; Toripalimab; Recombinant human endostatin (Endostar); Perioperative immunotherapy; PD-1 inhibitor; Anti-angiogenic therapy; Phase II study
MeSH Terms: conditions — Melanoma | interventions — endostar protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Arm (Experimental): Participants will:
  1. Receive 2 cycles of toripalimab before surgery (neoadjuvant therapy).
  2. Undergo surgical removal of the tumor.
  3. Post surgery, receive toripalimab every 2 weeks + Endostar (72-hour continuous infusion every 4 weeks) for up to 6 cycles (Endostar) or 11 cycles (toripalimab).
  4. Be monitored for tumor recurrence, side effects, and survival for up to 2 years after treatment.
  Interventions: Drug: Toripalimab combined with Endostar

INTERVENTIONS:
Drug: Toripalimab combined with Endostar — 1. Neoadjuvant Phase: 2 doses of toripalimab (240 mg IV, Q2W) before surgery.
  2. Surgery: Tumor resection within 2 weeks after the last neoadjuvant dose.
  3. Adjuvant Phase: 1) Toripalimab: 240 mg IV every 2 weeks (up to 11 cycles); 2) Endostar: 210 mg (72-hour continuous IV infusion) every 4 weeks (up to 6 cycles).

SUMMARY:
This is a Phase II clinical trial to evaluate the efficacy and safety of perioperative toripalimab (anti-PD-1) combined with recombinant human endostatin (Endostar) as postoperative adjuvant therapy in patients with clinical stage II cutaneous or acral malignant melanoma. The study aims to answer:

1. Does this combination improve the 2-year recurrence-free survival (2y-RFS) compared to historical data?
2. Is the treatment safe and tolerable for patients?

Participants will:

1. Receive 2 cycles of toripalimab before surgery (neoadjuvant therapy).
2. Undergo surgical removal of the tumor.
3. Post surgery, receive toripalimab every 2 weeks + Endostar (72-hour continuous infusion every 4 weeks) for up to 6 cycles (Endostar) or 11 cycles (toripalimab).
4. Be monitored for tumor recurrence, side effects, and survival for up to 2 years after treatment.

This is a single-arm, multicenter study involving 58 patients across several hospitals in China. Results will help determine if this combination could become a new standard adjuvant therapy for stage II melanoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, regardless of gender;
2. ECOG performance status: 0-1;
3. Patients with histologically or cytologically confirmed cutaneous or acral malignant melanoma, excluding mucosal and uveal melanoma;
4. Patients with BRAF, CKIT, and NRAS gene test results;
5. Treatment-naïve patients who have not received prior anti-tumor therapy;
6. Clinical stage II (AJCC 8th edition, 2017);
7. Laboratory tests must meet the following criteria:

   1. Hematology: Hemoglobin (Hb) ≥90 g/L (no transfusion within 14 days); absolute neutrophil count (ANC) ≥1.5×10^9/L; platelet count (PLT) ≥100×10^9/L;
   2. Biochemistry: Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×ULN; total bilirubin (TBIL) ≤1.5×ULN; serum creatinine (Cr) ≤1.5×ULN, and creatinine clearance >50 μmol/L;
   3. Coagulation: Activated partial thromboplastin time (APTT), international normalized ratio (INR), and prothrombin time (PT) ≤1.5×ULN;
   4. Doppler ultrasound assessment: Left ventricular ejection fraction (LVEF) ≥50%;
8. Female patients must agree to use contraception (e.g., intrauterine device [IUD], oral contraceptives, or condoms) during the study and for 6 months after study completion. A negative serum or urine pregnancy test within 7 days before enrollment is required, and patients must be non-lactating. Male patients must agree to use contraception during the study and for 6 months after study completion;
9. Patients must voluntarily participate in the study, sign the informed consent form, and demonstrate good compliance.

Exclusion Criteria:

1. History of allergic reactions to biological products;
2. Patients with prior or concurrent malignancies within 5 years (except cured basal cell carcinoma of skin or carcinoma in situ of cervix);
3. Any active autoimmune disease or history of autoimmune disorders (including but not limited to: autoimmune hepatitis, interstitial pneumonia, enteritis, vasculitis, nephritis; asthma requiring bronchodilators for medical intervention). Exceptions include: vitiligo, psoriasis, alopecia not requiring systemic therapy, well-controlled type I diabetes, or hypothyroidism with normal thyroid function on replacement therapy;
4. Requirement for immunosuppressive therapy using systemic or absorbable topical corticosteroids (equivalent to prednisone >10mg/day) within 2 weeks prior to first dose;
5. Any history or evidence of bleeding diathesis regardless of severity; grade ≥3 bleeding events per CTCAE v5.0 within 4 weeks prior to first dose; or presence of unhealed wounds, fractures, active gastrointestinal ulcers, ulcerative colitis, tumors with active bleeding, or other conditions deemed by investigators to potentially cause gastrointestinal hemorrhage or perforation;
6. Patients with severe and/or uncontrolled comorbidities including:

   1. Poorly controlled hypertension (SBP ≥150 mmHg or DBP ≥90 mmHg);
   2. Unstable angina, myocardial infarction, ≥grade 2 congestive heart failure, or arrhythmias requiring treatment (including QTc ≥480ms) within 6 months prior to first dose;
   3. Active or uncontrolled severe infections (≥grade 2 per CTCAE);
   4. Clinically significant liver disease including viral hepatitis (active HBV infection with HBV DNA >1×10³ copies/mL or >500 IU/mL; HCV infection with HCV RNA >1×10³ copies/mL or >100 IU/mL), decompensated liver disease, or chronic hepatitis requiring antiviral therapy;
   5. HIV-positive status;
   6. Poorly controlled diabetes (fasting glucose ≥grade 2 per CTCAE);
   7. Urinalysis showing proteinuria ≥++ with 24-hour urinary protein >1.0 g;
7. Administration of live vaccines within 4 weeks prior to treatment or anticipated need during study;
8. Other conditions deemed by investigators to potentially lead to premature study termination, including: severe comorbidities (including psychiatric disorders) requiring concomitant therapy, significant laboratory abnormalities, or social/family factors that may compromise patient safety or data/sample collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2029-03-30 (Estimated)

PRIMARY OUTCOMES:
2-year recurrence-free survival rate (2-year RFS rate) | From enrollment to the end of the 2nd year of follow-up

SECONDARY OUTCOMES:
1-year distant metastasis-free survival rate (1-year DMFS rate) | From enrollment to the end of the 1st year
Overall survival (OS) | Through study completion, an average of 3 years
1-year recurrence-free survival rate (1-year RFS rate) | From enrollment to the end of the 1st year
2-year distant metastasis-free survival rate (2-year DMFS rate) | From enrollment to the end of the 2nd year

CONTACTS AND LOCATIONS:
Overall Officials: Chunmeng Wang, Dr., Principal Investigator — Fudan University
Locations (4):
- China (4):
  - Department of Musculoskeletal Oncology, Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Cancer center, Shanghai 411 hospital, China RongTong Medical Healthcare Group Co.Ltd./411 Hospital, Shanghai University, Shanghai, Shanghai Municipality
  - Department of Surgical Oncology, Fudan University Shanghai Cancer Center Minhang Branch Hospital, Shanghai, Shanghai Municipality
  - Department of Oncology, Tongren Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided
Undecided yet.